CLINICAL TRIAL: NCT03552029
Title: A Phase 1 Study of Milademetan in Combination With Quizartinib in Subjects With FLT3-ITD Mutant Acute Myeloid Leukemia That Are Relapsed/Refractory, or Newly Diagnosed and Unfit for Intensive Chemotherapy
Brief Title: Milademetan Plus Quizartinib Combination Study in FLT3-ITD Mutant Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated based on a business decision by the Sponsor.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3032-A-U105
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Results first posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapsed/Refractory; Newly Diagnosed; Unfit for Chemotherapy; Positive for FLT3-ITD Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — quizartinib; milademetan

STUDY DESIGN:
Intervention Model Description: Part 1 Single Group 1 Arm, Part 2 Parallel, 2 Cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 - Quizartinib + Milademetan (Experimental): Participants with relapsed/refractory FLT3-ITD Mutant AML receive quizartinib + milademetan at increasing and/or decreasing doses and schedules
  Interventions: Drug: Quizartinib; Drug: Milademetan
- Part 2 - Cohort 1 (Experimental): Participants with relapsed/refractory FLT3-ITD Mutant AML receive the recommended dose of quizartinib + milademetan determined by Part 1
  Interventions: Drug: Quizartinib; Drug: Milademetan
- Part 2 - Cohort 2 (Experimental): Participants with newly diagnosed FLT3-ITD Mutant AML unfit for chemotherapy receive the recommended dose of quizartinib + milademetan determined by Part 1
  Interventions: Drug: Quizartinib; Drug: Milademetan

INTERVENTIONS:
Drug: Quizartinib — 20 or 30 mg tablets for oral administration
  Other Names: AC220; Vanflyta
Drug: Milademetan — 5, 20, 80 or 200 mg capsules for oral administration
  Other Names: DS-3032b
  Arms: Part 1 - Quizartinib + Milademetan
Drug: Milademetan — 5, 20, 80 or 200 mg capsules for oral administration; 30, 45, 80, or 100 mg capsules may be utilized
  Other Names: DS-3032b
  Arms: Part 2 - Cohort 1; Part 2 - Cohort 2

SUMMARY:
Participants with AML that have gone into remission and come back (relapsed) or gone into remission with a number of leukemia cells still in their system (refractory) will be recruited for this study. They will also be positive for FLT3-ITD mutation.

Participants will receive a combined dose of quizartinib and milademetan that have not been approved by the US Food and Drug Administration yet (m).

The combination of these drugs will be provided in different amounts on defined days (dosing schedules).

It is expected that the combination of milademetan and quizartinib will be safe and well tolerated. It is expected that the combination may fight the leukemia better than a single drug.

The study will run for approximately 3 years. There may be up to 156 participants.

The study has 2 parts:

* Part 1 will test 24-36 participants in approximately 15 study centers globally. Participants will receive two study drugs (milademetan and quizartinib) in different amounts on specific days. Information will be gathered to see what dosing schedule of the drug combination is best (maximum tolerated/recommended dose).
* Part 2 of the study will confirm the recommended dosing schedule identified in Part 1 is effective. A larger number of participants will receive the recommended dose in approximately 15 additional sites worldwide as necessary, based on the enrollment rate, the population, and the standard of care available to them at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Has reached ≥18 years old or the age of the age of majority in their country
* Part 1 (dose escalation): Has FLT3-ITD mutant (≥ 3% FLT3-ITD/total FLT3) AML (primary AML, secondary, or therapy-related AML), and has treatment failure to prior AML therapy or have relapsed after prior AML therapy
* Part 2 (dose expansion): Has FLT3-ITD mutant (≥3% FLT3-ITD/total FLT3) AML (primary, secondary, or therapy-related AML), and has treatment failure to prior AML therapy or have relapsed after prior AML therapy, OR has newly diagnosed AML who are ineligible for intensive induction chemotherapy
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (or 3 for patients with newly diagnosed AML between 18 and 74 years old)
* Has protocol-defined adequate renal, hepatic and cardiac status
* Is not pregnant, and if not postmenopausal or a surgically sterile male or female, is willing to use a highly effective contraceptive method upon enrollment, during the course of the study, and for 6 months following the last dose of investigational drug
* Is able and willing to provide protocol-defined bone marrow biopsies/aspirates

Exclusion Criteria:

* Has central nervous system (CNS) involvement of leukemia - patients with a history of CNS leukemia may be eligible if the CNS leukemia is adequately controlled (defined as no clinical symptoms of CNS disease and at least 2 consecutive lumbar punctures with no evidence of disease prior to study enrollment) after discussion and approval from the Sponsor
* Has acute promyelocytic leukemia (AML subtype M3)
* Has uncontrolled or significant cardiovascular disease or QTc interval >450 ms (average of triplicate determination)
* Has an uncontrolled infection requiring intravenous antibiotics, antivirals, or antifungals.
* Has known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection based on positive tests during Screening
* Has persistent, clinically significant > Grade 1 non-hematologic toxicity from prior AML therapies
* Has any history or medical condition, metastatic condition, drug/medication use or other condition that might, per protocol or in the opinion of the investigator, compromise:

  1. safety or well-being of the participant or offspring
  2. safety of study staff
  3. analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Daiichi Sankyo
Locations (8):
- United States (8):
  - Ronald Reagan Medical Center, UCLA, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Kansas Cancer Center, Fairway, Kansas
  - Rogel Cancer Center, University of Michigan, Ann Arbor, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke University Cancer Center, Durham, North Carolina
  - Sidney Kimmel Cancer Center, Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Zhang W, Li L, Muftuoglu M, Basyal M, Togashi N, Iwanaga K, Tanzawa F, Numata M, Bixby DL, Erba HP, Podoltsev N, Schiller GJ, Kumar P, Lesegretain A, Isoyama T, Seki T, Daver N, Andreeff M. Synergistic Activity of Combined FLT3-ITD and MDM2 Inhibition with Quizartinib and Milademetan in FLT3-ITD Mutant/TP53 Wild-type Acute Myeloid Leukemias. Clin Cancer Res. 2025 Jul 15;31(14):3033-3047. doi: 10.1158/1078-0432.CCR-24-2764. PMID 40327322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 out of the 22 screened participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 8 clinic sites in the United States. Only Part 1 is reported since the study terminated prior to Part 2.
Groups:
- Part 1, Cohort 1: Quizartinib + Milademetan: Participants with relapsed/refractory FLT3-ITD Mutant AML who received milademetan 90 mg daily (QD) Day 1 - Day 14 and quizartinib 30 mg QD.
- Part 1, Cohort 1A: Quizartinib + Milademetan: Participants with relapsed/refractory FLT3-ITD Mutant AML who received milademetan 90 mg daily (QD) Day 1 - Day 7 and quizartinib 30 mg QD.
Period: Overall Study
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan
Started | 4 | 6
Completed | 0 | 0
Not Completed | 4 | 6
Not completed — Death | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Enrolled Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Median (Full Range); unit: years] | 64 [51 to 72] | 65 [51 to 81] | 64 [51 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Following Administration of Milademetan in Combination With Quizartinib
Description: A dose limiting toxicity (DLT) is defined as any non-hematological treatment-emergent adverse event (TEAE) unless incontrovertibly related to disease progression, intercurrent illness, or concomitant medication, that occurs during the DLT evaluation period (28 days) in each dose level cohort, and is Grade 3 or higher according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, with exceptions specified: Grade 3 or higher aspartate aminotransferase (AST)/alanine aminotransferase (ALT) levels, OR elevation in total bilirubin ≥3.0 × upper limit of normal (ULN) that does not return to ≤Grade 2 elevation within 7 days. Absolute neutrophil count (ANC) <0.5 × 10^9/L, platelets <20 × 10^9/L, and marrow cellularity <5% at 6 weeks or later from start of therapy without any evidence of leukemia.
Time Frame: Baseline up to 28 days (Cycle 1) from the start of study drug administration
Population: Dose-limiting toxicities were assessed in the DLT Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan
Number analyzed (Participants) | 2 | 6
Participants | 1 | 0

2. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events by System Organ Class Following Administration of Milademetan in Combination With Quizartinib
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that emerges during the treatment period (from date of first dose up to 35 days after the last dose of the study treatment), having been absent at pretreatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment related to the pretreatment state, when the AE is continuous. AEs collected after 35 days after the last dose of study drug were not considered TEAEs unless they were treatment-related.
Time Frame: Baseline up to 35 days after last dose of study drug, up to approximately 2 years 3 months
Population: Treatment-emergent adverse events (irrespective of causality) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan
Number analyzed (Participants) | 4 | 6
Participants
  Any TEAEs | 4 | 6
  Any Blood and Lymphatic System Disorders | 2 | 5
  Any Cardiac Disorders | 1 | 2
  Any Ear and Labyrinth Disorders | 1 | 1
  Any Eye Disorders | 2 | 0
  Any Gastrointestinal Disorders | 4 | 6
  Any General Disorders and Administration Site Conditions | 3 | 5
  Any Immune System Disorders | 1 | 0
  Any Infections and Infestations | 4 | 1
  Any Injury, Poisoning and Procedural Complications | 0 | 3
  Any Investigations | 3 | 5
  Any Metabolism and Nutrition Disorders | 4 | 5
  Any Musculoskeletal and Connective Tissue Disorders | 2 | 4
  Any Nervous System Disorders | 4 | 3
  Any Psychiatric Disorders | 2 | 2
  Any Renal and Urinary Disorders | 1 | 2
  Any Respiratory, Thoracic, and Mediastinal Disorders | 4 | 4
  Any Skin and Subcutaneous Tissue Disorders | 3 | 5
  Any Vascular Disorders | 3 | 1

3. Secondary Outcome: Number of Participants With Best Overall Response Following Administration of Milademetan in Combination With Quizartinib
Description: Based on European LeukemiaNet criteria, complete remission (CR) was bone marrow (BM) blasts <5%, absence of circulating blasts/blasts with Auer rods, absence of extramedullary disease (EMD), absolute neutrophil count (ANC) ≥1.0×10^9/L, and platelet count ≥100×10^9/L; CR with Incomplete Blood Count Recovery (CRi): all CR criteria except for residual neutropenia or thrombocytopenia; Morphologic Leukemia Free State (MLFS): BM blasts <5%, absence of blasts with Auer rods, absence of EMD, and no hematologic recovery required; Partial Remission (PR): decrease of BM blast percentage by at least 50% (to 5% to 25%) and all criteria of CR; Stable disease: absence of CR, CRi, MLFS, or PR, and criteria for progressive disease (PD) not met; Relapse (after CR/CRi): BM blasts ≥5%, or reappearance of leukemic blasts, or EMD development; and PD: increase in BM blast % and/or increase of absolute blast counts: >50% increase in marrow blasts over baseline, >50% increase in peripheral blasts, or new EMD.
Time Frame: Baseline up to first documented response, disease progression, withdrawal, or death (whichever occurs first), up to approximately 2 years 3 months
Population: Best Overall Response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan
Number analyzed (Participants) | 4 | 6
Participants
  Complete remission (CR) | 0 | 0
  Complete Remission with Partial Hematological Recovery (CRh) | 0 | 0
  Complete Remission with Incomplete Blood Count Recovery (CRi) | 1 | 3
  Morphologic Leukemia Free State (MLFS) | 0 | 0
  Partial Remission (PR) | 0 | 0
  Stable Disease (SD) | 1 | 2
  Relapse | 0 | 0
  Missing | 2 | 1

4. Secondary Outcome: Overall Response Rate Following Administration of Milademetan in Combination With Quizartinib
Description: Overall response rate was defined as the number of participants with composite Complete Remission (CRc)+Morphological Leukemia Free State (MLFS)+Partial Remission (PR) based on the European LeukemiaNet criteria.
  Based on the European LeukemiaNet criteria, CRc was defined as complete remission (CR) as bone marrow (BM) blasts <5%, absence of circulating blasts/blasts with Auer rods, absence of extramedullary disease (EMD), absolute neutrophil count (ANC) ≥1.0×10^9/L, and platelet count ≥100×10^9/L; CR with Incomplete Blood Count Recovery (CRi): all CR criteria except for residual neutropenia or thrombocytopenia; Morphologic Leukemia Free State (MLFS): BM blasts <5%, absence of blasts with Auer rods, absence of EMD, and no hematologic recovery required; Partial Remission (PR): decrease of BM blast percentage by at least 50% (to 5% to 25%) and all criteria of CR.
Time Frame: as for outcome 3
Population: Overall response rate was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan
Number analyzed (Participants) | 4 | 6
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from date of first dose up to 35 days after last dose of study drug, up to approximately 2 years 3 months.
Description: A TEAE is defined as an adverse event (AE) that emerges during the treatment period (from date of first dose up to 35 days after the last dose of the study treatment), having been absent at pretreatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment related to the pretreatment state, when the AE is continuous.
Arm/Group | Part 1, Cohort 1: Quizartinib + Milademetan | Part 1, Cohort 1A: Quizartinib + Milademetan
All-Cause Mortality (participants affected / at risk) | 3/4 | 1/6
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1: Quizartinib + Milademetan (N=4) | Part 1, Cohort 1A: Quizartinib + Milademetan (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1: Quizartinib + Milademetan (N=4) | Part 1, Cohort 1A: Quizartinib + Milademetan (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Retinal exudates (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 4
Generalised oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 1
Swelling face (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2
Blood fibrinogen decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Fibrin D dimer increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Urine output decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Phonophobia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated based on a business decision by the Sponsor and was not due to a safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT03552029/Prot_SAP_000.pdf